CLINICAL TRIAL: NCT03796754
Title: Integration of the YoBEKA Program (Yoga, Movement, Relaxation, Concentration and Mindfulness) Into Elementary Schools in Germany
Brief Title: YoBEKA Program (Yoga, Movement, Relaxation, Concentration and Mindfulness) in Elementary Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: YoBEKA
Record Dates: First submitted 2019-01-02; First posted 2019-01-08 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YoBEKA Intervention (Active Comparator)
  Interventions: Behavioral: YoBEKA
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: YoBEKA — The teachers and students of the YoBEKA study arm receive a guided YoBEKA practice from an experienced YoBEKA trainer during the regular 4 month intervention period. The YoBEKA program is based on a combination of different, easy to perform exercises appropriate to the school situation, consisting of postures, verses for speech, song and movement, affirmations in movement to promote balance and coordination, and various rest and silence exercises to promote body awareness and relaxation techniques. The teaching is ideologically neutral and without religious background. The participating teachers receive an initial two-hour YoBEKA introductory course. Every 2 weeks there is a one to two-hour training course. The pedagogical specialists are supported once a week by an experienced YoBEKA trainer. The teachers are encouraged to integrate the learned exercises independently and regularly into their everyday school life.
  Arms: YoBEKA Intervention

SUMMARY:
The aim of this study is a first evaluation of the effectiveness of the YoBEKA Program (Yoga, Movement, Relaxation, Concentration and Mindfulness) to evaluate potential effects in stress reduction and concomitant psychological parameters.

ELIGIBILITY:
Inclusion criteria:

* Students from participating primary schools in Berlin aged 6-12 years
* Written declaration of consent of the parent or legal guardian

Exclusion criteria:

* Serious chronic or acute diseases
* Immobility or serious restriction for gymnastic exercises due to orthopaedic, neurological or other medical causes
* Participation in another study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Questionnaire on the assessment of stress and stress management in childhood and adolescence - Revision (SSKJ 3-8 R) | Change baseline, 4 months
  Filled out by students, assessing composite score (range 29-94): subscale 1 (stress-vulnerability [range 7-28]) summed with subscale 3 (stress symptoms and well-being [range 22-66]), lower score meaning a better outcome

SECONDARY OUTCOMES:
Inventory of the quality of life of children and adolescents (KIDSCREEN-27 children) | Change Baseline, 4 months, 12 months
  Filled out by students, assessing full scale, range 27-135, lower score meaning a better outcome
Perceived Stress Scale (PSS) | Change Baseline, 4 months, 12 months
  Filled out by teachers, assessing full scale, range 0-40, lower score meaning a better outcome
Teacher anxiety and stress inventory (LASI) | Change Baseline, 4 months, 12 months
  Filled out by teachers, assessing LASI 2, range 46-230, higher score meaning a better outcome
Screening for somatoform disorders of childhood and adolescence (SOMS-E) | Change Baseline, 4 months, 12 months
  Filled out by parents, assessing full scale, range 55-110, lower score meaning a better outcome
Inventory of the quality of life of children and adolescents (KIDSCREEN-52 parents) | Change Baseline, 4 months, 12 months
  Filled out by parents, assessing full scale, range 27-135, lower score meaning a better outcome

OTHER OUTCOMES:
Heart rate variability | Baseline, 4 months, 12 months
  Assessed with Faros 180 over 24 hours
Qualitative interviews | 4 months, 12 months
  Semi-structured interviews in focus groups

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University, Berlin, Germany